CLINICAL TRIAL: NCT00756834
Title: A Multi-center, Controlled, Consecutive Collection of Screening or Diagnostic Full Field Digital Mammography Images Acquired on the Mammomat Novation DR System for Development and Validation of Computer Aided Detection (CAD) Software
Brief Title: Case Collection Study for Collecting Images for the Development and Validation of Computer Aided Detection Software
Status: Terminated | Type: Observational
Why Stopped: No longer pursuing FDA submission/approval.
Sponsor: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: SMS-SP04-04
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Computer Aided Detection
MeSH Terms: conditions — Breast Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Mammography Image Collection: Acquired images
  Interventions: Device: Screening
- CAD Radiologist Reader: Retrospective reader study
  Interventions: Device: Screening

INTERVENTIONS:
Device: Screening — The MammoDetector™ Pro is a computer-aided software intended to identify and mark regions of interest on standard mammographic views to bring them to the attention of the radiologist after the initial reading has been completed. Thus, the device assists the radiologist in minimizing observational oversights by identifying areas on the original mammogram that may warrant a second review

SUMMARY:
The study objective is to assess the performance of the MammoDetector Pro to correctly mark biopsy-proven breast cancers imaged on the Siemens Mammomat Novation FFDM system compared to conventional film-screen mammography.

DETAILED DESCRIPTION:
The study design is a controlled study. The study is designed to demonstrate that the performance of the MammoDetector™ Pro on biopsy-proven malignant cases obtained with the Siemens Mammomat NovationDR FFDM system is not inferior to its performance on biopsy-proven malignant cases obtained with conventional film-screen mammography (FSM). The overall sensitivity of the MammoDetector™ Pro with both imaging modalities will be compared. Furthermore, the study is designed to demonstrate that the false marks noted by the MammoDetector™ Pro on routine screening "Normal" cases obtained with the FFDM system is not inferior those marked by the software on routine screening "Normal" cases obtained with conventional film-screen mammography (FSM).

ELIGIBILITY:
Inclusion Criteria:

1. Mammograms obtained from women 40 years of age and over;
2. Mammograms obtained from women only;
3. There are at least four standard views (right cranio-caudal [RCC], right medio-lateral oblique [RMLO], left cranio-caudal [LCC], left medio-lateral oblique [LMLO]) of the breast;
4. Informed consent is obtained.

   Mammograms of biopsy-proven cancer cases will be considered eligible for inclusion in the study if they meet the following criteria:
5. Biopsy-proven malignant case that was assigned a BI-RADS category 4 or 5 with a suspicious lesion and the corresponding pathology report for the suspicious lesion is available.
6. Cases which have one or more lesion.

   Routine screening "Normal" cases will be considered eligible for inclusion in the study if they meet the following criteria:
7. The case is a routine screening mammogram assigned a BI-RADS category 1 or 2 by a certified radiologist

Exclusion Criteria:

Cases are excluded from the study if they have any of the following conditions:

1. Mammographic needle projection or pre-biopsy markings are evident on the mammogram (these may cause false marks).
2. The mammograms include artifacts created by breast implant.
3. The mammograms are of poor quality (e.g., the digital image has very poor contrast);

   Mammograms of biopsy-proven cancer cases will be excluded from the study if they have any of the following conditions:
4. Cases in which the lesion is only palpable or visible by another modality (e.g., Ultrasound, MRI).
5. The pathology is not related to a specific region. That is, there is more than one biopsy region and the pathology reports cannot be related to the appropriate mammographic lesion. For example, a mammogram with multiple lesions and multiple related pathology reports on the same date and it is not clear which pathology report belongs to each lesion.
6. The pathology report is more than three months after the FFDM or FSM mammogram.
7. The mammogram was performed for the purpose of planning cancer therapy (e.g., radiation) (BIRADS 6).
8. Cases in which the lesion is characterized as an architectural distortion. -

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women 40 and older
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2006-11; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
The study will assess the performance of the MammoDetector™ Pro to correctly mark biopsy-proven breast cancers imaged on the Siemens Mammomat NovationDR FFDM system compared to conventional film-screen mammography (FSM). | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Louise Ebbert, Study Director — Siemens Medical Solutions
Locations (1):
- Siemens Medical Solutions, Malvern, Pennsylvania, United States